CLINICAL TRIAL: NCT06441292
Title: Study on Prostate Targeted Biopsy Precision Navigation Method Based on Multi-Modal Image Fusion Deep Learning Using Multi-Parameter Ultrasound and MRI
Brief Title: Multi-Modal Image Fusion for Precision Prostate Biopsy Navigation
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai East Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: PB-NAV-MMIF-01
Record Dates: First submitted 2024-05-28; First posted 2024-06-04 (Actual); Last update posted 2024-06-04 (Actual); Status verified 2024-05

CONDITIONS: Prostate Cancer
Keywords: Prostate Cancer; targeted biopsy
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- conventional biopsy group (Active Comparator): undergo standard prostate biopsy procedures without additional technological assistance
  Interventions: Procedure: Non-AI-assisted
- AI-assisted biopsy group (Experimental): utilize advanced deep learning models that integrate multi-modal image fusion from multi-parameter ultrasound and MRI to guide the biopsy process
  Interventions: Procedure: AI-assisted

INTERVENTIONS:
Procedure: AI-assisted — utilize advanced deep learning models that integrate multi-modal image fusion from multi-parameter ultrasound and MRI to guide the biopsy process
  Arms: AI-assisted biopsy group
Procedure: Non-AI-assisted — undergo standard prostate biopsy procedures without additional technological assistance
  Arms: conventional biopsy group

SUMMARY:
This study is a prospective randomized controlled clinical trial aimed at comparing the detection rates of clinically significant prostate cancer between conventional biopsy methods and AI-assisted biopsy methods in patients undergoing initial prostate biopsy who meet the indications for prostate biopsy.

DETAILED DESCRIPTION:
This study is a prospective randomized controlled clinical trial designed to investigate the efficacy of AI-assisted biopsy methods compared to conventional biopsy methods in detecting clinically significant prostate cancer. The target population includes patients undergoing their initial prostate biopsy who meet established indications for prostate biopsy.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 18
2. PSA > 4 ng/ml and/or abnormal DRE
3. Sign the informed consent

Exclusion Criteria:

1. Have acute or chronic prostatitis
2. Contraindications to prostate biopsy
3. Contraindications to MRI
4. Other reasons that not suitable for this trial

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 602 (Estimated)
Dates: Start 2024-07-01 (Estimated); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-07-15 (Estimated)

PRIMARY OUTCOMES:
The detection rate of clinically significant prostate cancer by targeted biopsy alone | 2-3 weeks post-biopsy
  The proportion of men with a Gleason score ≥3+4 in pathological assessment for targeted biopsy samples

SECONDARY OUTCOMES:
The detection rate of clinically significant prostate cancer by targeted biopsy combined with template biopsy | 2-3 weeks post-biopsy
  The proportion of men with a Gleason score ≥3+4 in pathological assessment for combined targeted biopsy samples
The detection rate of any prostate cancer by targeted biopsy alone | 2-3 weeks post-biopsy
  The proportion of men with a Gleason score ≥3+3 in pathological assessment for targeted biopsy samples
The detection rate of any prostate cancer by targeted biopsy combined with template biopsy | 2-3 weeks post-biopsy
  The proportion of men with a Gleason score ≥3+3 in pathological assessment for combined targeted biopsy samples

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai East Hospital, Tongji University School of Medicine, Shanghai, China

IPD SHARING:
Plan to Share IPD: No